CLINICAL TRIAL: NCT05389735
Title: Evaluation of Ventilation Distribution With Electrical Impedance Tomography in Mechanically Ventilated Patients After Surgery: a Prospective Observational Study
Brief Title: Evaluation of Postoperative Ventilation Distribution With Electrical Impedance Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: hi38655072
Record Dates: First submitted 2022-05-15; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Electrical Impedance Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative patients require respiratory management . It is known that the intrapulmonary ventilation distribution becomes uneven due to dorsal atelectasis and ventral hyperinflation during mechanical ventilation management, but the incidence in postoperative patients is unknown. EIT is a device that can monitor the ventilation distribution in the lungs over time without being exposed to the bedside. Therefore, for patients at risk of postoperative respiratory complications, use EIT to 1) evaluate the pulmonary ventilation distribution during postoperative ventilation management, 2) pulmonary ventilation distribution and postoperative respiratory organs. The purpose of this study is to clarify the relationship with the severity of complications.

A prospective observational study to investigate the relationship between ventilation distribution and prognosis using EIT in patients undergoing mechanical ventilation after adult surgery.

ELIGIBILITY:
1. Patients aged 18 years or older who have undergone surgery
2. Patients undergoing mechanical ventilation management when returning to the ICU after surgery
3. High-risk patients with postoperative respiratory complications

Exclusion Criteria:

1. the EIT belt is worn Patients with unstable spine or pelvis due to fractures, etc. Patients with implantable defibrillation and implantable pacemaker Patients with skin lesions such as blisters between the 4th and 5th intercostal spaces where
2. Patients with DNR (do-not-resuscitate)
3. Patients undergoing home ventilator management before surgery
4. Preoperative, hypocardiac function patients (echocardiography shows left ventricular ejection fraction of 40% or less, or NYHA III degree or more +)
5. Patients with a ventricular assist device
6. Patients with extracorporeal membrane oxygenation (VV or VA)
7. History of neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postoperative patients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Association the dorsal fraction of ventilation in EIT and postoperative respiratory complication score | up to 12 weeks
  Dorsal fraction of ventilation(%):The dorsal fraction of ventilation is calculated as the sum of all pixel values in the dorsal half of the EIT image over the sum of all pixel values from the EIT image
  Postoperative pulmonary complications score(0-5):Postoperative pulmonary complications were scored using a grade scale ranging from 0 to 5, with grade zero representing absence of complications, grades 1 to 4 representing increasing (worsening) levels of complications, and grade 5 representing death before hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Osaka University, Osaka, Japan